CLINICAL TRIAL: NCT02371226
Title: A Phase 1 Safety and Dose-Finding Study of a Human Insulin Receptor Monoclonal Antibody-Human Alpha-L-iduronidase (HIRMAb-IDUA) Fusion Protein, AGT-181 in Adult Patients With Mucopolysaccharidosis I (MPS I, Hurler Syndrome)
Brief Title: Safety and Dose Ranging Study of Insulin Receptor MAb-IDUA Fusion Protein in Patients With MPS I
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ArmaGen, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGT-181-102
Record Dates: First submitted 2015-02-19; First posted 2015-02-25 (Estimated); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Mucopolysaccharidosis I
Keywords: MPS I
MeSH Terms: conditions — Mucopolysaccharidosis I | interventions — valanafusp alpha

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Experimental): 1 mg/kg AGT-181 (fusion protein of anti-human insulin receptor monoclonal antibody and alpha-L-iduronidase; HIRMAb-IDUA) administered once weekly x 8 weeks
  Interventions: Drug: AGT-181 (HIRMAb-IDUA)
- Cohort 2 (Experimental): 3 mg/kg AGT-181 (HIRMAb-IDUA) administered once weekly x 8 weeks
  Interventions: Drug: AGT-181 (HIRMAb-IDUA)
- Cohort 3 (Experimental): 6-9 mg/kg AGT-181 (HIRMAb-IDUA) administered once weekly x 8 weeks
  Interventions: Drug: AGT-181 (HIRMAb-IDUA)

INTERVENTIONS:
Drug: AGT-181 (HIRMAb-IDUA) — intravenous infusion over 3-4 hours
  Other Names: fusion protein of monoclonal antibody to human insulin receptor fused to alpha-L-iduronidase

SUMMARY:
AGT-181 is a fusion protein containing alpha-L-Iduronidase that is intended to deliver the enzyme peripherally and to the brain, when administered intravenously. This study is a safety and dose ranging study to obtain safety and exposure data, as well as information on the biological activity of the investigational drug.

ELIGIBILITY:
Inclusion Criteria:

* Male age 18 years or older
* Diagnosis of MPS I (documented fibroblast or leukocyte IDUA enzyme activity level of less than 10% of the lower limit of the normal range of the measuring laboratory)
* Voluntary written consent by patient or legally responsible representative
* All women of childbearing potential and sexually mature males must be advised to use a medically accepted method of contraception throughout the study.
* Negative pregnancy test (females)
* Must not have received ERT for at least 6 weeks prior to AGT-181 treatment
* Must have elevated urinary GAGs if no ERT has been received in the prior 3 months

Exclusion Criteria:

* Refusal to complete baseline evaluations.
* Any medical condition or other circumstances that may significantly interfere with study compliance
* Receipt of an investigational drug within the prior 90 days
* History of diabetes mellitus or hypoglycemia
* Clinically significant spinal cord compression, evidence of cervical instability.
* Known hypersensitivity to alpha-L-iduronidase or any of the components of AGT-181.
* Known to be nonresponsive to standard ERT treatment.
* Previously successful (engrafted) hematopoietic stem cell transplantation that resulted in normalization of urinary GAGs.
* Contraindication for lumbar puncture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-01-23 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | eight weeks

SECONDARY OUTCOMES:
plasma pharmacokinetic parameters (maximal concentration, half-life, area under the curve, mean residence time, volume of distribution and clearance of AGT-181) | 8 weeks
change in urinary or plasma glycosaminoglycans (GAGs) | 8 weeks
change in liver size | 8 weeks
change in spleen size | 8 weeks
change in levels of heparan sulfate and dermatan sulfate in the cerebrospinal fluid | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Rioux, MD PhD, Study Director — ArmaGen, Inc
Locations (6):
- United States (6):
  - Children's Hospital Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Emory Healthcare, Decatur, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - University of Utah Hospital, Salt Lake City, Utah